CLINICAL TRIAL: NCT06488521
Title: A Single-blind Randomized Comparative Study of the Safety and Pharmacokinetics of Complarate and Actemra® in the Form of a Solution for Subcutaneous Administration in Parallel Groups of Healthy Volunteers
Brief Title: A Safety and Pharmacokinetics Study of Complarate (Tocilizumab Biosimilar Solution) and Actemra® in Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GNR087s-RA012
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: tocilizumab; humanized monoclonal antibodies; safety; pharmacokinetics; equivalence; biosimilar; IL-6 receptor; solution; subcutaneous administration
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complarate (JSC "GENERIUM", Russia) (Experimental): tocilizumab biosimilar
  Interventions: Biological: Complarate
- Actemra® (F. Hoffmann-La Roche Ltd., Switzerland) (Active Comparator): tocilizumab
  Interventions: Biological: Actemra®

INTERVENTIONS:
Biological: Complarate — Complarate solution, a subcutaneous injection at a single dose of 162 mg.
  Other Names: Tocilizumab biosimilar
  Arms: Complarate (JSC "GENERIUM", Russia)
Biological: Actemra® — Actemra® solution, subcutaneous injection at a single dose of 162 mg.
  Other Names: Tocilizumab
  Arms: Actemra® (F. Hoffmann-La Roche Ltd., Switzerland)

SUMMARY:
This is a randomized single-blind comparative parallel group study of the safety, pharmacokinetics of the solution form of Complarate and Actemra® in healthy volunteers. Participants received a single subcutaneous dose of tocilizumab 162 mg. The follow up period was 43 days.

DETAILED DESCRIPTION:
Complarate (tocilizumab, solution) is being developed as a biosimilar to the drug Actemra®, a solution for subcutaneous injection.

Tocilizumab is a recombinant humanized monoclonal antibody to the human interleukin-6 (IL-6) receptor from the immunoglobulin G1 (IgG1) subclass. Tocilizumab binds to and inhibits both soluble and membrane IL-6 receptors (sIL-6R and mIL-6R).

This I phase study is aimed to compare the pharmacokinetics and safety of the drugs Complarate and Actemra® after their single subcutaneous administration to healthy volunteers at a dose of 162 mg. The study included healthy volunteers aged 18-45 years at the time of signing the informed consent form. The study included a screening period, single administration of study/comparator drug and a follow up period. Allocation of patients to treatment groups was carried out by randomization in a ratio of 1:1 to the study drug and comparator drug. 256 patients (128 to the study drug group and 128 to the comparator drug group) are being randomized.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study;
* Men and women aged 18 to 45 years, inclusive, at the time of signing the informed consent form;
* Verified diagnosis "healthy" (based on a detailed medical history, in the absence of deviations from normal values during a physical examination, assessment of vital signs, as well as according to laboratory tests, electrocardiography and digital fluorography/digital pulmonary radiography);
* Body weight from 50.0 to 90.0 kg, inclusive; body mass index from 18.5 to 29.9 kg/m2, inclusive;
* Volunteer's agreement to adhere to adequate methods of contraception for 3 months after administration of the study or reference drug;
* The volunteer's consent not to become a donor of blood and/or its components during the entire study and for 30 days after its completion.

Exclusion Criteria:

* Hypersensitivity to any of the components of the study or reference drug; a history of allergic reactions requiring drug treatment;
* Any history of tocilizumab use; use of tumor necrosis factor-alfa (TNF-alpha) inhibitors less than 3 months before randomization;
* The presence of acute and chronic diseases of the cardiovascular system, respiratory system, nervous, immune and endocrine systems, gastrointestinal tract, liver and biliary tract, kidneys and urinary tract, blood and lymphatic system, mental illness, tuberculosis;
* History of an autoimmune disease;
* History of cancer;
* Acute infectious diseases that resolved less than 28 days before randomization;
* Use of prescription medications less than 28 days or 5 half-lives of the drug (whichever is longer) or systematic use of over-the-counter medications/dietary supplements less than 14 days before randomization;
* Blood donation or blood loss (450 ml of blood or more) less than 3 months before randomization and/or planned blood donation in any quantity during participation in the study;
* Participation in clinical trials of medicinal products less than 3 months or 5 half-lives of the study drug (whichever is longer) before randomization in this study;
* Regular alcohol consumption exceeding 5 units. alcohol per week (where each unit is equal to 30 ml of ethyl alcohol) or information about a history of alcoholism, drug addiction, or drug abuse;
* Positive test for the presence of alcohol in exhaled air;
* Positive urine test for the content of narcotic and potent drugs;
* Positive test for hepatitis B or C, HIV or syphilis;
* Any surgical interventions planned during the period of participation in the study;
* Depot injections or use of implants of any other drugs less than 3 months before randomization;
* Immunization with any vaccine less than 3 months before randomization;
* Special lifestyle (work at night);
* Pregnancy or breastfeeding period;
* Unwillingness or inability to comply with the recommendations prescribed by this protocol;
* Other reasons that, in the opinion of the investigator and/or Sponsor, prevent the volunteer from participating in the study or create an unreasonable risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) | Day 43
  Analysis of equivalence of area under concentration-time curve from time 0 (predose) to the last quantifiable data point and to infinity of Complarate and Actemra®
Pharmacokinetics: Peak Plasma Concentration (Cmax) | Day 43
  Analysis of equivalence of Cmax of Complarate and Actemra®

SECONDARY OUTCOMES:
Proportion of volunteers with adverse events (AE) | Day 43
  The Investigator will carefully monitor each subject throughout the study for any adverse events (coded to preferred term and system organ class using the Medical Dictionary for Regulatory Activities [MedDRA])
Proportion of volunteers with ADA | Day 43
  Antidrug antibodies (ADA) level

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — JSC GENERIUM
Locations (3):
- Russia (3):
  - State budgetary healthcare institution of the city of Moscow "City Clinic No. 2 of the Moscow Health Department", Moscow, Moscow
  - Federal State Autonomous Educational Institution of Higher Education First Moscow State Medical University named after I.M. Sechenov Ministry of Health of Russia, Moscow, Moscow
  - LLC "X Seven Clinical Research", Saint Petersburg, Sankt-Peterburg

IPD SHARING:
Plan to Share IPD: No